CLINICAL TRIAL: NCT06806670
Title: Effects of Exercise and Dietary Counselling in Reducing the Cardiovascular Risk Score in Kidney Transplant Patients: KT- LIFESTYLE Study
Brief Title: Exercise and Diet Effects in Reducing Cardiovascular Risk in Kidney Transplant Recipients
Acronym: KT-LIFESTYLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: CNT (Centro Nazionale Trapianti) (Unknown); Azienda Unità Sanitaria Locale della Romagna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KT LIFESTYLE; RC24000854 - 2790615 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-11-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-07

CONDITIONS: Kidney Transplant Recipients
Keywords: exercise; diet; cardiovascular risk; kidney transplant recipients; gut microbiota; lifestyle
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A, lifestyle intervention (Experimental): lifestyle intervention
  Interventions: Behavioral: lifestyle intervention
- Group B (No Intervention): standard of care

INTERVENTIONS:
Behavioral: lifestyle intervention — exercise and dietary counselling
  Arms: Group A, lifestyle intervention

SUMMARY:
The goal of this clinical trial is to assess whether, over an observation period of 3 years, there is a reduction in cardiovascular risk, and the extent of this reduction, in a group of adult kidney transplant patients undergoing tailored exercise combined with dietary counselling compared to a group of patients following the 'standard of care'.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

* Prescribed exercise and dietary counselling could reduce of at least 1% in the cardiovascular risk score (by Framingham score) and cardiovascular biomarkers in kidney transplant recipients?
* How much can a lifestyle intervention affect kidney function, quality of life and the gut microbiota in this patient population?

Researchers will compare kidney transplant recipients undergoing tailored exercise combined with dietary counselling compared to a group of patients following the 'standard of care' to see if there is a reduction in cardiovascular risk, BMI, inflammatory markers, improve of gut microbiota and perception of quality of life. In addition, a number of hospital admissions for important clinical events, the number of fatal and non-fatal cardiovascular events (MACE), and mortality from all causes will be assessed in the long term.

Participants will enroll from the Nephrology, Dialysis and Transplant Units and randomize in intervantion group (A) or control (B).

In group A/intervention, a tailored exercise programme combined with specific dietary counselling will be prescribed, in group B/control, generic advice on healthy lifestyles will be given (standard of care) without specific prescription.

In all patients, quality of life, gut microbiota, inflammatory and cardiovascular biomarkers (Framingham score, BNP, etc.), lipid profile and renal function over time will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stabilised male and female kidney transplant patients (assessment by the referring transplant centre)
* Minimum age, 30 years;
* Maximum age, 69 years;
* Period since transplantation: from 6 months (subject to clinical stability being achieved) to 10 years;
* Organ function: eGFR (CKD-EPI formula) ≥ 30 mL/min/1.73m ;2
* Obtaining informed consent;

Exclusion Criteria:

* Patients unable to follow the prescription,
* Recent acute cardiovascular event (< 2 months),
* Unstable angina,
* Hyperkinetic/hypokinetic arrhythmias not controlled by therapy, and with signs of haemodynamic impairment,
* Severe aortic stenosis,
* Heart failure NYHA class III-IV, FE < 40%,
* Acute illnesses that limit physical activity,
* Severe hypertension (basal BP ≥200/110 mm Hg),
* Neuro-musculo-skeletal pathologies that may be aggravated by exercise,
* Patients unwilling to change lifestyle;
* Any form of substance abuse, psychiatric disorder or condition that, according to the investigator, can complicate communication between doctor and patient;
* Pregnant women.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular risk reduction | From enrollment to the end of the treatment (3 years)
  reduction of at least 1% in the cardiovascular risk score - Framingham score - over the observation time. This score estimates the risk of developing a cardiovascular event over a 10-year period and is calculated in relation to the outcome from the following identifiable variables in normal clinical practice:
  * Sex
  * Age
  * Systolic pressure value
  * Treatment for hypertension (yes/no)
  * Smoker (yes/no)
  * Diabetes (yes/no)
  * HDL value
  * Total cholesterol value

SECONDARY OUTCOMES:
Renal function | From enrollment to the end of the treatment (3 years)
  The trend of renal function assess by eGFR using the CKD-EPI formula
Gut microbiota analysis | From enrollment to the end of the treatment (3 years)
  The relative abundances of the main intestinal bacterial groups and hence the effect of physical exercise on the gut microbiota
Inflammatory status | From enrollment to the end of the treatment (3 years)
  The variation of the inflammatory status (by CRP analysis, IL-6, ferritin, cortisol)
Quality of Life (QoL) | From enrollment to the end of the treatment (3 years)
  The perception of quality of life through the SF12 questionnaire (composite items of physical and mental health)
Adherence to the lifestyle intervention | From enrollment to the end of the treatment (3 years)
  Adherence to dedicated counseling through IPAQ questionnaire to assess physical activity and food frequency questionnaire to assess diet
Cost-effectiveness of a healthy lifestyle intervention | From enrollment to the end of the treatment (3 years)
  number of hospital admissions for major clinical events
Cardiovascular biomarkers | From enrollment to the end of the treatment (3 years)
  the trend of biomarkers related to cardiovascular risk (lipid profile, BNP)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Tarantino, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Padua Netto MV, Bonfim TC, Costa EN, de Lima HV, Netto LC. Cardiovascular risk estimated in renal transplant recipients with the Framingham score. Transplant Proc. 2012 Oct;44(8):2337-40. doi: 10.1016/j.transproceed.2012.07.054. PMID 23026587
- [Background] Henry RM, Kostense PJ, Bos G, Dekker JM, Nijpels G, Heine RJ, Bouter LM, Stehouwer CD. Mild renal insufficiency is associated with increased cardiovascular mortality: The Hoorn Study. Kidney Int. 2002 Oct;62(4):1402-7. doi: 10.1111/j.1523-1755.2002.kid571.x. PMID 12234312
- [Background] Sarnak MJ, Levey AS, Schoolwerth AC, Coresh J, Culleton B, Hamm LL, McCullough PA, Kasiske BL, Kelepouris E, Klag MJ, Parfrey P, Pfeffer M, Raij L, Spinosa DJ, Wilson PW; American Heart Association Councils on Kidney in Cardiovascular Disease, High Blood Pressure Research, Clinical Cardiology, and Epidemiology and Prevention. Kidney disease as a risk factor for development of cardiovascular disease: a statement from the American Heart Association Councils on Kidney in Cardiovascular Disease, High Blood Pressure Research, Clinical Cardiology, and Epidemiology and Prevention. Hypertension. 2003 Nov;42(5):1050-65. doi: 10.1161/01.HYP.0000102971.85504.7c. No abstract available. PMID 14604997
- [Background] Totti V, Fernhall B, Di Michele R, Todeschini P, La Manna G, Cappuccilli M, Angelini ML, De Fabritiis M, Merni F, Benedetti E, Roi GS, Nanni Costa A, Mosconi G. Longitudinal Analysis of Cardiovascular Risk Factors in Active and Sedentary Kidney Transplant Recipients. Medicina (Kaunas). 2020 Apr 16;56(4):183. doi: 10.3390/medicina56040183. PMID 32316125
- [Background] Masiero L, Puoti F, Bellis L, Lombardini L, Totti V, Angelini ML, Spazzoli A, Nanni Costa A, Cardillo M, Sella G, Mosconi G. Physical activity and renal function in the Italian kidney transplant population. Ren Fail. 2020 Nov 10;42(1):1192-1204. doi: 10.1080/0886022X.2020.1847723. PMID 33256487
- [Background] Totti V, Tame M, Burra P, Mosconi G, Roi GS, Sella G, Ermolao A, Ferrarese A, Sgarzi S, Savino G, Parodi G, Poggioli G, Ricchiuti A, Di Michele R, Trerotola M, Nanni Costa A. Physical Condition, Glycemia, Liver Function, and Quality of Life in Liver Transplant Recipients After a 12-Month Supervised Exercise Program. Transplant Proc. 2019 Nov;51(9):2952-2957. doi: 10.1016/j.transproceed.2019.03.087. Epub 2019 Oct 10. PMID 31607623
- [Background] Roi GS, Mosconi G, Totti V, Angelini ML, Brugin E, Sarto P, Merlo L, Sgarzi S, Stancari M, Todeschini P, La Manna G, Ermolao A, Tripi F, Andreoli L, Sella G, Anedda A, Stefani L, Galanti G, Di Michele R, Merni F, Trerotola M, Storani D, Nanni Costa A. Renal function and physical fitness after 12-mo supervised training in kidney transplant recipients. World J Transplant. 2018 Feb 24;8(1):13-22. doi: 10.5500/wjt.v8.i1.13. PMID 29507858
- [Background] Kohl HW 3rd, Craig CL, Lambert EV, Inoue S, Alkandari JR, Leetongin G, Kahlmeier S; Lancet Physical Activity Series Working Group. The pandemic of physical inactivity: global action for public health. Lancet. 2012 Jul 21;380(9838):294-305. doi: 10.1016/S0140-6736(12)60898-8. PMID 22818941
- [Background] van der Ploeg HP, Bull FC. Invest in physical activity to protect and promote health: the 2020 WHO guidelines on physical activity and sedentary behaviour. Int J Behav Nutr Phys Act. 2020 Nov 26;17(1):145. doi: 10.1186/s12966-020-01051-1. PMID 33239047
- [Background] Markell MS, Armenti V, Danovitch G, Sumrani N. Hyperlipidemia and glucose intolerance in the post-renal transplant patient. J Am Soc Nephrol. 1994 Feb;4(8 Suppl):S37-47. doi: 10.1681/ASN.V48s37. PMID 8193294
- [Background] Painter P. Exercise following organ transplantation: A critical part of the routine post transplant care. Ann Transplant. 2005;10(4):28-30. PMID 17037085
- [Background] Seoane-Pillado MT, Pita-Fernandez S, Valdes-Canedo F, Seijo-Bestilleiro R, Pertega-Diaz S, Fernandez-Rivera C, Alonso-Hernandez A, Gonzalez-Martin C, Balboa-Barreiro V. Incidence of cardiovascular events and associated risk factors in kidney transplant patients: a competing risks survival analysis. BMC Cardiovasc Disord. 2017 Mar 7;17(1):72. doi: 10.1186/s12872-017-0505-6. PMID 28270107
- [Background] Lim WH, Lok C, Kim SJ, Knoll G, Shah B, Naylor K, McArthur E, Luo B, Dixon SN, Hawley C, Ooi E, Viecelli AK, Wong G. Incidence of Major Adverse Cardiovascular Events and Cardiac Mortality in High-Risk Kidney-Only and Simultaneous Pancreas-Kidney Transplant Recipients. Kidney Int Rep. 2021 Feb 23;6(5):1423-1428. doi: 10.1016/j.ekir.2021.02.019. eCollection 2021 May. No abstract available. PMID 34013120
- [Background] Regolisti G, Maggiore U, Sabatino A, Gandolfini I, Pioli S, Torino C, Aucella F, Cupisti A, Pistolesi V, Capitanini A, Caloro G, Gregorini M, Battaglia Y, Mandreoli M, Dani L, Mosconi G, Bellizzi V, Di Iorio BR, Conti P, Fiaccadori E; Gruppo di Studio "Esercizio fisico nel paziente con insufficienza renale cronica" of the Societa Italiana di Nefrologia. Correction: Interaction of healthcare staff's attitude with barriers to physical activity in hemodialysis patients: A quantitative assessment. PLoS One. 2018 Jun 20;13(6):e0198987. doi: 10.1371/journal.pone.0198987. eCollection 2018. PMID 29924872
- [Background] Pang A, Lingham S, Zhao W, Leduc S, Rakel A, Sapir-Pichhadze R, Mathur S, Janaudis-Ferreira T. Physician Practice Patterns and Barriers to Counselling on Physical Activity in Solid Organ Transplant Recipients. Ann Transplant. 2018 May 22;23:345-359. doi: 10.12659/AOT.908629. PMID 29784902